CLINICAL TRIAL: NCT05922397
Title: Evaluation of Clinical Outcomes and Acceptability of an Anatomical Classification for Placenta Accreta Spectrum, a Multicentric Prospective Cohort Study
Brief Title: Placenta Accreta Spectrum Topographic Classification
Status: Recruiting | Type: Observational
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Other Study IDs: FVL-2125
Record Dates: First submitted 2023-05-31; First posted 2023-06-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-07

CONDITIONS: Placenta Accreta
Keywords: Pregnancy outcomes; Topographic classification; Placenta accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study is a prospective multicenter study consisting of a cohort of patients with prenatal or intraoperative diagnosis of PAS, evaluating the clinical outcomes of the group of patients found in each category of the topographic classification. In addition, an approach to evaluate the acceptability of this classification among the obstetrician-gynecologists of the participating medical centers will be included.

DETAILED DESCRIPTION:
The aim of this study is to describe the demographic and clinical characteristics of patients with a diagnosis of placenta accreta spectrum, and to determine the correlation between the topographic classification and the clinical outcomes found in the study. Finally, to evaluated whether the proposed classification is accepted by the obstetrician-gynecologists of the participating centers that manage placenta accreta spectrum patients.

It is an observational, multicentric study of a prospective cohort, in which data will be obtained from the medical records and other documents in each participating center, which are considered to be of routine use in day-to-day clinical practice. The study of the outcomes proposed in this protocol will be limited to those recorded in the clinical records and will be taken into account until the participant is discharged from the hospital, during which a surgical intervention was performed due to the suspicion or diagnosis of PAS.

It is projected that the period of patient enrollment will last 2 years, counting on from the first participant included. The study population is pregnant patients with a diagnosis of placenta accreta spectrum who visits any of the participating medical centers, and also obstetrician-gynecologists working in participating medical centers.

The centers invited to participate are hospitals or clinics that already have knowledge in how to apply the surgical staging of PAS, and the topographic classification and have experience using it.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman over 18 years old.
* Prenatal diagnosis by ultrasound or MRI of Placenta Accreta Spectrum (PAS), regardless of the suspected degree of severity of the disease.
* Case requiring surgical management, either as scheduled or emergent procedure.
* Application of the topographic classification of placenta accreta spectrum during laparotomy.

Exclusion Criteria:

* None.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Pregnant patients with a diagnosis of placenta accreta spectrum who visits any of the participating medical centers.
  * Obstetrician-gynecologists working in participating medical centers.
Sampling Method: Probability Sample
Enrollment: 326 (Estimated)
Dates: Start 2023-05-21 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Days of postoperative hospitalization | From the day the surgery is performed until the day of discharge or the date of death from any cause, whichever occurs first, evaluated up to 42 days.
  Number of days the patient was hospitalized from the day of surgery to the day of discharge
Volume of intraoperative blood loss | During surgery
  Surgical bleeding calculated in milliliters
Bladder injury | Up to 42 days postpartum
  Number of patients who had Bladder injuries
Surgical reintervention | Up to 42 days postpartum
  Number of patients who need surgical reoperation after index surgery
Complications associated with vascular interventions | Up to 42 days postpartum
  The patient presented thrombosis or other complication during post-surgery associated with vascular interventions.
Maternal death | 24 months
  Does the patient die during this study

CONTACTS AND LOCATIONS:
Overall Officials: Albaro J Nieto-Calvache, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundación Valle del Lili, Cali, Colombia

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data, since we are not allowed to share information concerning the medical history of our patients or health workers

REFERENCES:
- [Background] Palacios-Jaraquemada JM, Fiorillo A, Hamer J, Martinez M, Bruno C. Placenta accreta spectrum: a hysterectomy can be prevented in almost 80% of cases using a resective-reconstructive technique. J Matern Fetal Neonatal Med. 2022 Jan;35(2):275-282. doi: 10.1080/14767058.2020.1716715. Epub 2020 Jan 26. PMID 31984808
- [Background] Kingdom JC, Hobson SR, Murji A, Allen L, Windrim RC, Lockhart E, Collins SL, Soleymani Majd H, Alazzam M, Naaisa F, Shamshirsaz AA, Belfort MA, Fox KA. Minimizing surgical blood loss at cesarean hysterectomy for placenta previa with evidence of placenta increta or placenta percreta: the state of play in 2020. Am J Obstet Gynecol. 2020 Sep;223(3):322-329. doi: 10.1016/j.ajog.2020.01.044. Epub 2020 Jan 30. PMID 32007492
- [Background] Palacios-Jaraquemada JM, D'Antonio F. Possible limitation to use the International Federation of Gynecology and Obstetrics classification of placenta accreta spectrum. Am J Obstet Gynecol. 2020 Dec;223(6):944. doi: 10.1016/j.ajog.2020.06.033. Epub 2020 Jun 19. No abstract available. PMID 32565238
- [Background] Nieto-Calvache AJ, Palacios-Jaraquemada JM, Aryananda RA, Rodriguez F, Ordonez CA, Messa Bryon A, Calvache JPB, Lopez J, Campos CI, Mejia M, Rengifo M, Galliadi LMV, Maya J, Zambrano MA, Aguayo IP, Carabali IG, Burgos JM. How to identify patients who require aortic vascular control in placenta accreta spectrum disorders? Am J Obstet Gynecol MFM. 2022 Jan;4(1):100498. doi: 10.1016/j.ajogmf.2021.100498. Epub 2021 Oct 2. PMID 34610485
- [Background] Jauniaux E, Jurkovic D, Hussein AM, Burton GJ. New insights into the etiopathology of placenta accreta spectrum. Am J Obstet Gynecol. 2022 Sep;227(3):384-391. doi: 10.1016/j.ajog.2022.02.038. Epub 2022 Mar 3. PMID 35248577
- [Background] Garmi G, Salim R. Epidemiology, etiology, diagnosis, and management of placenta accreta. Obstet Gynecol Int. 2012;2012:873929. doi: 10.1155/2012/873929. Epub 2012 May 7. PMID 22645616
- [Background] Jauniaux E, Ayres-de-Campos D, Langhoff-Roos J, Fox KA, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO classification for the clinical diagnosis of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2019 Jul;146(1):20-24. doi: 10.1002/ijgo.12761. PMID 31173360
- [Background] Collins SL, Stevenson GN, Al-Khan A, Illsley NP, Impey L, Pappas L, Zamudio S. Three-Dimensional Power Doppler Ultrasonography for Diagnosing Abnormally Invasive Placenta and Quantifying the Risk. Obstet Gynecol. 2015 Sep;126(3):645-653. doi: 10.1097/AOG.0000000000000962. PMID 26214694
- [Background] Hussein AM, Elbarmelgy RA, Elbarmelgy RM, Thabet MM, Jauniaux E. Prospective evaluation of impact of post-Cesarean section uterine scarring in perinatal diagnosis of placenta accreta spectrum disorder. Ultrasound Obstet Gynecol. 2022 Apr;59(4):474-482. doi: 10.1002/uog.23732. Epub 2022 Mar 8. PMID 34225385
- [Background] Allen L, Jauniaux E, Hobson S, Papillon-Smith J, Belfort MA; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Nonconservative surgical management. Int J Gynaecol Obstet. 2018 Mar;140(3):281-290. doi: 10.1002/ijgo.12409. No abstract available. PMID 29405317
- [Background] Sentilhes L, Kayem G, Chandraharan E, Palacios-Jaraquemada J, Jauniaux E; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Conservative management. Int J Gynaecol Obstet. 2018 Mar;140(3):291-298. doi: 10.1002/ijgo.12410. No abstract available. PMID 29405320
- [Background] Melber DJ, Berman ZT, Jacobs MB, Picel AC, Conturie CL, Zhang-Rutledge K, Binder PS, Eskander RN, Roberts AC, McHale MT, Ramos GA, Ballas J, Kelly TF. Placenta Accreta Spectrum Treatment With Intraoperative Multivessel Embolization: the PASTIME protocol. Am J Obstet Gynecol. 2021 Oct;225(4):442.e1-442.e10. doi: 10.1016/j.ajog.2021.07.001. Epub 2021 Jul 7. PMID 34245679
- [Background] Shamshirsaz AA, Fox KA, Erfani H, Clark SL, Salmanian B, Baker BW, Coburn M, Shamshirsaz AA, Bateni ZH, Espinoza J, Nassr AA, Popek EJ, Hui SK, Teruya J, Tung CS, Jones JA, Rac M, Dildy GA, Belfort MA. Multidisciplinary team learning in the management of the morbidly adherent placenta: outcome improvements over time. Am J Obstet Gynecol. 2017 Jun;216(6):612.e1-612.e5. doi: 10.1016/j.ajog.2017.02.016. Epub 2017 Feb 16. PMID 28213059
- [Background] Hussein AM, Kamel A, Raslan A, Dakhly DMR, Abdelhafeez A, Nabil M, Momtaz M. Modified cesarean hysterectomy technique for management of cases of placenta increta and percreta at a tertiary referral hospital in Egypt. Arch Gynecol Obstet. 2019 Mar;299(3):695-702. doi: 10.1007/s00404-018-5027-7. Epub 2019 Jan 4. PMID 30607590
- [Background] Sentilhes L, Seco A, Azria E, Beucher G, Bonnet MP, Branger B, Carbillon L, Chiesa C, Crenn-Hebert C, Dreyfus M, Dupont C, Fresson J, Huissoud C, Langer B, Morel O, Patrier S, Perrotin F, Raynal P, Rozenberg P, Rudigoz RC, Vendittelli F, Winer N, Deneux-Tharaux C, Kayem G; PACCRETA Study Group. Conservative management or cesarean hysterectomy for placenta accreta spectrum: the PACCRETA prospective study. Am J Obstet Gynecol. 2022 Jun;226(6):839.e1-839.e24. doi: 10.1016/j.ajog.2021.12.013. Epub 2021 Dec 14. PMID 34914894
- [Background] Whittington JR, Pagan ME, Nevil BD, Kalkwarf KJ, Sharawi NE, Hughes DS, Sandlin AT. Risk of vascular complications in prophylactic compared to emergent resuscitative endovascular balloon occlusion of the aorta (REBOA) in the management of placenta accreta spectrum. J Matern Fetal Neonatal Med. 2022 Aug;35(16):3049-3052. doi: 10.1080/14767058.2020.1802717. Epub 2020 Aug 11. PMID 32781879
- [Background] Nieto-Calvache AJ, Hidalgo-Cardona A, Lopez-Giron MC, Rodriguez F, Ordonez C, Garcia AF, Mejia M, Pabon-Parra MG, Burgos-Luna JM. Arterial thrombosis after REBOA use in placenta accreta spectrum: a case series. J Matern Fetal Neonatal Med. 2022 Nov;35(21):4031-4034. doi: 10.1080/14767058.2020.1846178. Epub 2020 Nov 18. PMID 33207992
- [Background] Chandraharan E. Need for an urgent paradigms shift in thinking to avoid serious maternal morbidity and mortality associated with PAS. Best Pract Res Clin Obstet Gynaecol. 2021 Apr;72:1-3. doi: 10.1016/j.bpobgyn.2021.04.001. No abstract available. PMID 33894905
- [Background] Aryananda RA, Aditiawarman A, Gumilar KE, Wardhana MP, Akbar MIA, Cininta N, Ernawati E, Wicaksono B, Joewono HT, Dachlan EG, Bachtiar CA, Kurniawati D, Virdayanti DP, Ariani G, Dekker GA, Sulistyono A. Uterine conservative-resective surgery for selected placenta accreta spectrum cases: Surgical-vascular control methods. Acta Obstet Gynecol Scand. 2022 Jun;101(6):639-648. doi: 10.1111/aogs.14348. Epub 2022 Mar 17. PMID 35301710
- [Background] Palacios Jaraquemada JM, Garcia Monaco R, Barbosa NE, Ferle L, Iriarte H, Conesa HA. Lower uterine blood supply: extrauterine anastomotic system and its application in surgical devascularization techniques. Acta Obstet Gynecol Scand. 2007;86(2):228-34. doi: 10.1080/00016340601089875. PMID 17364288
- [Background] Nieto-Calvache AJ, Palacios-Jaraquemada JM, Aryananda R, Basanta N, Aguilera R, Benavides JP, Lopez J, Campos C, Valencia L, Arboleda K, Cabrera V, Cabrera J, Tavera-Martinez GM, Sinisterra S, Maya J, Pena T, Burgos-Luna JM, Messa A. How to perform the one-step conservative surgery for placenta accreta spectrum move by move. Am J Obstet Gynecol MFM. 2023 Feb;5(2):100802. doi: 10.1016/j.ajogmf.2022.100802. Epub 2022 Nov 11. PMID 36372188
- [Background] Sargent W, Collins SL. Are women antenatally diagnosed with abnormally invasive placenta receiving optimal management in England? An observational study of planned place of delivery. Acta Obstet Gynecol Scand. 2019 Mar;98(3):337-341. doi: 10.1111/aogs.13487. Epub 2018 Nov 15. PMID 30368768
- [Background] Brown AD, Hart JM, Modest AM, Hess PE, Abbas AM, Nieto-Calvache AJ, Bhide A, Lim B, Dunjin C, Palacios-Jaraquemada J, Sentilhes L, Soma-Pillay P, Aryananda RA, Hantoushzadeh S, Wang S, Shamshirsaz AA, Shainker SA. Geographic variation in management of patients with placenta accreta spectrum: An international survey of experts (GPASS). Int J Gynaecol Obstet. 2022 Jul;158(1):129-136. doi: 10.1002/ijgo.13960. Epub 2021 Oct 28. PMID 34610154
- [Background] Nieto-Calvache AJ, Lopez-Giron MC, Nieto-Calvache A, Messa-Bryon A, Benavides-Calvache JP, Burgos-Luna JM. A nationwide survey of centers with multidisciplinary teams for placenta accreta patient care in Colombia, observational study. J Matern Fetal Neonatal Med. 2022 Jun;35(12):2331-2337. doi: 10.1080/14767058.2020.1786052. Epub 2020 Jul 6. PMID 32627610
- [Background] Nieto-Calvache AJ, Palacios-Jaraquemada JM, Hidalgo A, Vergara-Galliadi LM, Cortes Charry R, Aguilera Daga LR, Verastegui Goyzueta R, Osanan G, Fernandez J, Corrales F, Mereci W, Yuen-Chon V, Guevara E, Zuniga LA, Giron, Turcios FE, Munoz H, Perez AM, Meade P, Basanta N, Pineda JP. Management practices for placenta accreta spectrum patients: a Latin American hospital survey. J Matern Fetal Neonatal Med. 2022 Dec;35(25):6104-6111. doi: 10.1080/14767058.2021.1906858. Epub 2021 Apr 11. PMID 33843408
- [Background] Nieto AJ, Echavarria MP, Carvajal JA, Messa A, Burgos JM, Ordonez C, Benavidez JP, Mejia M, Lopez L, Fernandez PA, Escobar MF. Placenta accreta: importance of a multidisciplinary approach in the Colombian hospital setting. J Matern Fetal Neonatal Med. 2020 Apr;33(8):1321-1329. doi: 10.1080/14767058.2018.1517328. Epub 2018 Sep 25. PMID 30153754
- [Background] Einerson BD, Watt MH, Sartori B, Silver R, Rothwell E. Lived experiences of patients with placenta accreta spectrum in Utah: a qualitative study of semi-structured interviews. BMJ Open. 2021 Nov 3;11(11):e052766. doi: 10.1136/bmjopen-2021-052766. PMID 34732490
- [Background] Nieto-Calvache AJ, Palacios-Jaraquemada JM, Aguilera LR, Arriaga W, Colonia A, Aryananda RA, Nieto-Calvache AS, Maya J, Vergara-Galliadi LM, Messa Bryon A. Telemedicine facilitates surgical training in placenta accreta spectrum. Int J Gynaecol Obstet. 2022 Jul;158(1):137-144. doi: 10.1002/ijgo.14000. Epub 2021 Nov 20. PMID 34714947

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05922397/Prot_SAP_000.pdf